CLINICAL TRIAL: NCT05767515
Title: The Effects of Acetyl L--Carnitine and Myo/Chiro-Inositol on Improving Ovulation, Pregnancy Rate, Ovarian Function and Perceived Stress Response in Patients With PCOS
Brief Title: The Effects of Acetyl-L-Carnitine and Myo/Chiro-Inositol in Patients With PCOS
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Collaborators: University of Cagliari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NO:KMU/IBMS/2020/45; F.No.SG-21-153/RDC/691 (Other Grant/Funding Number: NIH,Pakistan)
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Infertility, Female; PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
Keywords: PCOS, INFERTILTY
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome | interventions — Metformin; Inositol; Acetylcarnitine

STUDY DESIGN:
Intervention Model Description: Treatment of PCOS with Myo/D-chiro Inositol and comparison with metformin
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metformin Group (Active Comparator): Metformin will be used in dose of 1000 mg BD daily for 30 infertile female PCOS patients
  Interventions: Drug: metformin
- Inositol isomers Group (Experimental): Inositols isomers (Myo inositol and D- Chiro Inositol in its physiological ratio) will be used 2000mg BD Daily for 30 infertile female PCOS patients
  Interventions: Drug: metformin
- Acetyl-L- Carnitine Group (Experimental): Acetyl-L-Carnitine will be given in dose of 1000mgBD Daily for 30 infertile female PCOS patients
  Interventions: Drug: metformin
- Combine Group (Experimental): Inositol isomers and Acetyl-L-Carnitine will be given in dose of 2000mg and 1000mg respectively BD daily for 30 infertile female PCOS patients
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — Treatment of infertile female with PCOS with inositol isomers and Acetyl-L-Carnitine
  Other Names: myo inositol, D- chiro Inositol, Acetyl-L-Carnitine

SUMMARY:
The large number of women in their child bearing age is affected by Polycystic ovarian syndrome (PCOS) leading to infertility. However it is considered as a multisystem disorder with comorbidities rather than a gynecological and a dermatological problem. Patient mostly have anovulation presented as oligomennorhea or amenorrhea and hyperandrogenism presented as hirsutism along with hyperinsulinemia and insulin resistance. Many etiological factors are reported but those actually responsible for PCOS in females still need to be explored. However hyperandrogenism and insulin resistance being the key triggering condition apart from cardiovascular disease, type 2 diabetes, hypertension and obesity. World Health Organization (WHO) has considered Infertility's as public health problem. Researchers reported the obesity role in occurrence of PCOS and its Infertility's relation .

PCOS is not a simple pathophysiologic process for which one treatment address all manifestation. Treatment should target specific manifestations and individualized patient goals. First-line agents for ovulation induction and treatment of infertility in patients with PCOS include metformin and clomiphene alone or in combination. It has been approved as category "A "to regulate ovulation and improves pregnancy rates in women with PCOS . Mostly it result in complication like multiple follicle recruitment rate, multiple pregnancy and thinning of endometrial wall leading to early abortion and endometrial cancers. The use of naturally occurring compounds like myoinositol, D-chiro- inositol and L- carnitine which are already part of human body are expected to produce significant results without any side effects . The proposed study will provide an alternative to current treatments available for infertility due to PCOS. The expected project execution time is 2 years. Thus, the present project will discover new insights about treatment of infertility and thus generate new knowledge which will help Academia, scientists and health care professionals. Results of the study will be disseminated on different forums including to policy makers , Pharmaceutical, national and international agencies. The result will be published in journal both national and international with good impact factors. The outcome of the project will be used as publication in high impact international journals, filling of patents and will also be presented in national and international forums.

DETAILED DESCRIPTION:
Introduction A tremendously high number of women in their child bearing age is affected by Polycystic ovarian syndrome (PCOS) leading to infertility (1). PCOS is not a simple gynecological or dermatological problem but a multisystem disorder with comorbidities. Patients mostly have anovulation presented as oligomennorhea or amenorrhea and hyperandrogenism presented with symptoms of hirsutism along with hyperinsulinemia and insulin resistance. The presence of multiple cysts in the ovaries however, is not essential for diagnosis (2). Hyperandrogenism and insulin resistance being the key triggering condition apart from cardiovascular disease, type 2 diabetes, hypertension and obesity. PCOS and infertility involves genetic and environmental factors, however, in Pakistani the cultural background of intermarriages is contributing noticeably towards the multiplicity of disease (3). World Health Organization (WHO) has considered infertility as public health problem. It was the objective of UN conference 2015 to provide access and quality reproductive health services to all individuals. Management of PCOS require prolong use of pharmaceuticals which has serious effects sometimes even fatal, therefore the natural, easily available, cost effective nutraceuticals has tremendous effects and have now used safely in many clinical trials(4) The current study aims to provide evidence to support the use of neutraceuticals in the management of PCOS in infertile patients and their comparison with standard drug used in treatment of infertility caused by PCOS.. This study can help run a long way in achieving the millennium goals MDG(3) SGD(3) to which Pakistan is a signatory and to reduce maternal mortality and improve reproductive health of its female population The following agent is used as standard drug in an infertile women with PCOS in a clinical set-up Metformin a biguanide, used as first line drug for the treatment of diabetes and PCOS. It works by preventing hepatic gluconeogenesis and intestinal glucose absorption thus improving insulin sensitivity (5). In addition to its systemic effects on insulin signaling it effect autocrine/paracrine signaling in ovarian tissue thus improving ovarian steriodogensis and endometrial receptivity (6). In a recent study its role in infertile PCOS women was established resulting in significant number of ovulation and live birth than controls (7).

Complementary and alternative medicine approach for the treatment of PCOS is becoming popular in recent years. It is claimed that dietary supplements and herbal remedies are safer than conventional drugs.

Acetyl L-Carnitine : Carnitine a quaternary ammonium compound made in the body from lysine and methionine and is available in an active ( L) and an inactive (D ) form. L-carnitine is available in supplemental form and has significant role in enhancing metabolism, producing energy and protecting against oxidative stress. Role of carnitine in treating insulin resistance is being frequently discussed with reference to accrual of acyl-CoA derivatives (8). Hence as suggested if the normal levels of carnitine in the diabetics and obese patients is ensured the insulin insensitivity can be drastically improved. Further the level of L-carnitine in PCOS patients was found to be considerably less. Follicogensis is a highly energy dependent process on mitochondria. In PCOS the functioning of mitochondria is effected due to inflammation and other deregulations because of accumulation of testosterone and insulin in ovary. It help in transport of lipids from cytosol to mitochondria in breakdown of lipids for production of energy (9) Inositol; Inositols present in plants and animal a member of sugar alcohol comprising nine cyclohexane-1, 2, 3, 4, 5, 6-hexol stereoisomers. Being vitamin like it is made in human body as well as synthetically. It is a component of cell membrane and acts as a second messenger, has important role in release of different autacoids, hormones, and neurotransmitters (10).The promising role of two of its isomers namely Myo-inositol (MI) and D-chiro-inositol (DCI) in the treatment of PCOS has been documented. Studies have demonstrated that performance of MI to induce ovulation in patients with infertility due to PCOS can be improved if DCI is combined to it. Best results are achieved when the two isomers are used in 40:1 ratio which is the normal amount in which they exist in the body (11). Both MI and DCI can influence oxidative and non-oxidative metabolism. Apart from being involved in activation of multiple enzymes MI is involved in glucose transport and DCI in insulin production from B- cells and ATP production (12) DCI contributes in mediating insulin activity mainly on non-ovarian tissues, MI displays specific effects on ovary, chiefly by modulating glucose metabolism and FSH-signaling. Moreover, MI may also improve ovarian functions by modulating steroid metabolism through non-insulin-dependent pathways In PCOS patient due IR there is dysregulation in MI/DCI ratio in non- ovarian tissue related to reduced epimarse activity. However ovaries being insulin sensitive have lower level of MI than DCI due to increase epimerase activity (13).

Rationale The incidence of PCOS is increasing throughout the world. It is much higher in Pakistani women (52%) than Caucasian women (20-25%) and is contributing towards both primary (50%) and secondary (25%) infertility (14). Infertilty has its sociocultural connotations resulting in emotional and mental stress. Infertilty due to PCOS should be treated with nutraceuticals for being natural, cost effective, easily available and with minimum side effects. The inositol isomers in its physiological ratio (40:1) and carnitine as an antioxidant has shown significant effects in regularization of metabolic and endocrine parameters of the body Rationale of the present study is that Inositol and Carnitine alone and in combination may be a better alternate for treatment of infertility in patients with PCOS, compared to Metformin. To the best of our knowledge no study till date is documented for synergistic effects of Acetyl-L Carnitine and inositol isomers when used, in physiological balanced ratio, for infertilty Objectives 1. To compare the effects of Inositol isomers and Acetyl-LCarnitine ( alone and in combination) with Metformin on improving ovulation, pregnancy rate, restoring ovarian function, metabolic balance and perceived stress response in patient with PCOS Hypothesis It is hypothesized that Inositol and Acetyl L-Carnitine alone may produce better or at least comparable results to Metformin in improving Pregnancy rate, ovulation, restoring ovarian function, metabolic balance and perceived stress response in infertile patients with PCOS.

It is also hypothesized that the synergistic action of Inositol isomers and Acetyl L-Carnitine in combination may produce better or at least comparable results to Metformin in improving pregnancy rate, ovulation, restoring ovarian function, metabolic balance and perceived stress response in infertile patients with PCOS STUDY DESIGN: This will be a noncommercial randomized double blind clinical trial (RCT) in which subject and treatment provider will blinded to treatment intervention. In this study we will compare the treatment of naturally occurring nutraceuticals with Metformin (control group) which is used as first line drug in treatment of PCOS for infertile women. The nature of study will be explained in both Pashto and Urdu and informed consent will be taken SETTINHS: OPD patients in Gynecology and Obstetrics Department, Pakistan Institute of Medical Sciences, Islamabad (PIMS) and Bacha Khan Medical Complex, Swabi, (BKMC) KP DURATION: The study is expected to be completed in 1.year with duration for 6 months.

SAMPLE SIZE: The study will include 120 patients with PCOS according to our inclusion of the NIH 2012 extension of ESHRE/ASRM 2003 criteria.

.

ELIGIBILITY:
Inclusion Criteria:Married women with PCOS aged ≥18 years to ≤35 years who is infertile (primary and secondary) and have a wish to conceive will be included in the study. The diagnosis of PCOS will be made according to the NIH 2012 extension of ESHRE/ASRM 2003 criteria (21). Identiﬁcation of speciﬁc phenotypes will be included:

A. Hyperandrogenism plus Ovulatory dysfunction plus Polycystic Ovarian Morphology (HA +OD+PCOM) B. Hyperandrogenism plus Ovulatory dysfunction (HA+OD) C. Hyperandrogenism plus Poly Cystic Ovarian Morphology (HA+PCOM). D. Ovulatory dysfunction plus Polycystic Ovarian Morphology (OD+PCO)

Couple inclusion criteria; Being a sterility trial couples ensuing to do their semen analysis regularly or provide record showing their sperm concentration to be at least 15 million /ml in at least one ejaculation during the past one year with some motile sperm. Similarly, couples having ability and readiness to perform sexual intercourse as and when directed by the investigator will be included. Female subjects should have at least one open fallopian tube and normal uterus from inside on hysterosalpingography /hysteroscopy/laparoscopy or have normal course of conception, delivery during the past 03 years. Patients should have no history of tubal ligation or vasectomy procedure that has been reversed

Exclusion Criteria: Females having history of having an infertile male partner in the past, Cushing syndrome, diabetes, thyroid disorders, hyperprolactinemia, ovarian tumors, congenital adrenal hyperplasia, androgen-producing tumors, history of seizures, pregnancy undiagnosed vaginal bleeding History of suspected cervical or endometrial carcinoma breast carcinoma using contraceptive anti-coagulants, antiplatelet, isoproterenol and potassium sparing diuretics, anti-depressants and medications that alters the biochemical or hormonal profile will be excluded. Participants who have been prescribed hormones during the past at least 3 months before the study will not be included in the study. Patient who is willing to participate in the study is using any medicine that can be discontinued (e.g., oral contraceptive or ovulation induction agents (GnRH agonist and antagonist; gonadotropins, HCG) will be allowed wash out period of 02 months before being included in the study.

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertilty
Enrollment: 120 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
CLINICAL PREGNANCY | 6 MONTHS
  intrauterine pregnancy with positive fetal heart motion as determined on transvaginal ultrasound or HCG level is more than 1500IU/L

SECONDARY OUTCOMES:
OVULATION | 6 MONTHS
  will be defined as serum Progesterone ( ≥3ng/ml or 9.54nmol/l) r on u/s examination
Conception | 6 Months
  positive serum level of HCG
Biochemical Pregnancy | 6 months
  Falling B-HCG concentration on serial determination
tetosterone levels | 6 MONTHS
  clinically on mFG , Biochemically on FAI

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Medical University, Peshawar, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubin KH, Glintborg D, Nybo M, Abrahamsen B, Andersen M. Development and Risk Factors of Type 2 Diabetes in a Nationwide Population of Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3848-3857. doi: 10.1210/jc.2017-01354. PMID 28938447
- [Background] Orio F, Palomba S. Reproductive endocrinology: New guidelines for the diagnosis and treatment of PCOS. Nat Rev Endocrinol. 2014 Mar;10(3):130-2. doi: 10.1038/nrendo.2013.248. Epub 2013 Dec 10. PMID 24322653
- [Background] Akram M, Roohi N. Endocrine correlates of polycystic ovary syndrome in Pakistani women. J Coll Physicians Surg Pak. 2015 Jan;25(1):22-6. PMID 25604364
- [Background] Chauhan B, Kumar G, Kalam N, Ansari SH. Current concepts and prospects of herbal nutraceutical: A review. J Adv Pharm Technol Res. 2013 Jan;4(1):4-8. doi: 10.4103/2231-4040.107494. PMID 23662276
- [Background] An H, He L. Current understanding of metformin effect on the control of hyperglycemia in diabetes. J Endocrinol. 2016 Mar;228(3):R97-106. doi: 10.1530/JOE-15-0447. Epub 2016 Jan 7. PMID 26743209
- [Background] Mansfield R, Galea R, Brincat M, Hole D, Mason H. Metformin has direct effects on human ovarian steroidogenesis. Fertil Steril. 2003 Apr;79(4):956-62. doi: 10.1016/s0015-0282(02)04925-7. PMID 12749437
- [Background] Morley LC, Tang T, Yasmin E, Norman RJ, Balen AH. Insulin-sensitising drugs (metformin, rosiglitazone, pioglitazone, D-chiro-inositol) for women with polycystic ovary syndrome, oligo amenorrhoea and subfertility. Cochrane Database Syst Rev. 2017 Nov 29;11(11):CD003053. doi: 10.1002/14651858.CD003053.pub6. PMID 29183107
- [Background] Tauqir S, Israr M, Rauf B, Malik MO, Habib SH, Shah FA, Usman M, Raza MA, Shah I, Badshah H, Ehtesham E, Shah M. Acetyl-L-Carnitine Ameliorates Metabolic and Endocrine Alterations in Women with PCOS: A Double-Blind Randomized Clinical Trial. Adv Ther. 2021 Jul;38(7):3842-3856. doi: 10.1007/s12325-021-01789-5. Epub 2021 May 28. PMID 34047916
- [Background] Salehpour S, Nazari L, Hoseini S, Moghaddam PB, Gachkar L. Effects of L-carnitine on Polycystic Ovary Syndrome. JBRA Assist Reprod. 2019 Oct 14;23(4):392-395. doi: 10.5935/1518-0557.20190033. PMID 31294953
- [Background] 10. Porcaro G, Bizzarri M, Monastra G, et al Strategies for the treatment of polycystic ovary syndrome (PCOS) women: the role of myoinositol (MI) and d-chiro-inositol (DCI) between diet and therapy. Nova science publishers. 2016 1-18
- [Background] 11. Facchinetti F, Dante G, Neri I. The ratio of MI to DCI and its impact in the treatment of polycystic ovary syndrome: experimental and literature evidences. Front Gynecol Endocrinol 2015;3:103-9.
- [Background] Heimark D, McAllister J, Larner J. Decreased myo-inositol to chiro-inositol (M/C) ratios and increased M/C epimerase activity in PCOS theca cells demonstrate increased insulin sensitivity compared to controls. Endocr J. 2014;61(2):111-7. doi: 10.1507/endocrj.ej13-0423. Epub 2013 Nov 2. PMID 24189751
- [Background] Bevilacqua A, Bizzarri M. Inositols in Insulin Signaling and Glucose Metabolism. Int J Endocrinol. 2018 Nov 25;2018:1968450. doi: 10.1155/2018/1968450. eCollection 2018. PMID 30595691
- [Derived] Gul M, Khan H, Rauf B, Bukhari SMS, Ehtesham E, Malik MO, Shah FA, Alanazi FE, Shah M. Comparative efficacy of combined myo-inositol and D-chiro inositol versus metformin across PCOS Phenotypes: enhancing ovarian function, ovulation, and stress response in a prospective clinical trial. Naunyn Schmiedebergs Arch Pharmacol. 2025 Jul;398(7):8761-8772. doi: 10.1007/s00210-025-03813-9. Epub 2025 Jan 23. PMID 39847053